CLINICAL TRIAL: NCT00025597
Title: European Infant Neuroblastoma Study - Unresectable Tumors (MYCN Not Amplified)
Brief Title: Combination Chemotherapy Followed by Surgery in Treating Infants With Newly Diagnosed Neuroblastoma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Infant Neuroblastoma Study Group - 1999 (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068977; EURO-INF-NB-STUDY-1999-99.1; EU-20125A
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2001-11

CONDITIONS: Neuroblastoma
Keywords: localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: vincristine sulfate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by surgery in treating infants who have newly diagnosed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the survival and morbidity of infants with newly diagnosed stage II or III unresectable neuroblastoma without MYCN amplification treated with vincristine and cyclophosphamide, etoposide and carboplatin, and cyclophosphamide, doxorubicin, and vincristine followed by surgery.
* Determine whether deletion of chromosome 1p or diploidy/tetraploidy are prognostic factors in these patients.
* Determine whether there are other prognostic criteria that could be used in future therapeutic stratification of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to symptomatic spinal cord involvement (yes vs no).

Patients without evidence of symptomatic spinal cord compression receive vincristine IV on day 1 and cyclophosphamide IV on days 1-5. Treatment repeats every 14 days for 2 courses. Patients eligible for surgery undergo surgical resection and then are removed from the study.

Patients ineligible for surgery after 2 courses of initial chemotherapy, but with at least 25% response to initial chemotherapy, receive 2 additional courses of vincristine and cyclophosphamide. Patients eligible for surgery undergo surgical resection and then are removed from the study.

Patients ineligible for surgery after 2 additional courses of initial chemotherapy or with disease progression receive etoposide IV over 2 hours and carboplatin IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses. Patients eligible for surgery undergo surgical resection and then are removed from the study.

Patients who remain ineligible for surgery or with disease progression after etoposide and carboplatin receive cyclophosphamide IV over 1 hour on days 1-5, doxorubicin IV over 6 hours on days 4 and 5, and vincristine IV on days 1 and 5. Treatment repeats every 21 days for 2 courses. Patients then undergo surgical resection or biopsy.

Patients with symptomatic spinal cord compression receive initial treatment with etoposide and carboplatin as above. Patients with improved symptoms and resectable disease after initial chemotherapy undergo surgical resection or biopsy. Patients who remain ineligible for surgery or with no improvement in symptoms after initial chemotherapy receive cyclophosphamide, doxorubicin, and vincristine as above. Patients then undergo surgical resection or biopsy.

Patients are followed within 6 months and then annually for 5 years.

PROJECTED ACCRUAL: A total of 100 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed newly diagnosed stage II or III neuroblastoma or ganglioneuroblastoma

  * Unresectable disease
* No MYCN amplification (i.e., fewer than 10 copies)
* No metastases to bone marrow
* No radiological bone lesions in skeleton

PATIENT CHARACTERISTICS:

Age:

* Under 12 months at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No evidence of liver disease by ultrasound

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-07; Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Rubie, MD, Study Chair — Centre Hospitalier Regional de Purpan
Locations (11):
- St. Anna Children's Hospital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Centre Hospitalier Regional de Purpan, Toulouse, France
- Istituto Giannina Gaslini, Genoa, Italy
- Rikshospitalet University Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- Hospital Universitario LA FE, Valencia, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Bristol Royal Hospital for Children, Bristol, England, United Kingdom

REFERENCES:
- [Result] Rubie H, De Bernardi B, Gerrard M, Canete A, Ladenstein R, Couturier J, Ambros P, Munzer C, Pearson AD, Garaventa A, Brock P, Castel V, Valteau-Couanet D, Holmes K, Di Cataldo A, Brichard B, Mosseri V, Marquez C, Plantaz D, Boni L, Michon J. Excellent outcome with reduced treatment in infants with nonmetastatic and unresectable neuroblastoma without MYCN amplification: results of the prospective INES 99.1. J Clin Oncol. 2011 Feb 1;29(4):449-55. doi: 10.1200/JCO.2010.29.5196. Epub 2010 Dec 20. PMID 21172879